CLINICAL TRIAL: NCT06379386
Title: Long-term Prognosis and Valve Durability of Transcatheter Aortic Valve Replacement for Aortic Valve Disease: a Real-world, Prospective, Single-center, Observational Study
Brief Title: Long-term Prognosis and Valve Durability of TAVR
Status: Recruiting | Type: Observational
Sponsor: Xijing Hospital (Other)
Responsible Party: Principal Investigator, LingTao, Professor in Cardiology, Director of the department of Cardiology, Xijing Hospital
Other Study IDs: TRACE TAVR Registry
Record Dates: First submitted 2024-04-18; First posted 2024-04-23 (Actual); Last update posted 2024-04-23 (Actual); Status verified 2024-04

CONDITIONS: Aortic Valve Stenosis and Insufficiency
Keywords: Aortic Valve Disease; TAVR; Prognosis; Valve durability
MeSH Terms: conditions — Aortic Valve Stenosis; Aortic Valve Disease | interventions — Transcatheter Aortic Valve Replacement

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Procedure: Transcatheter aortic valve replacement — A total of 1000 consecutive patients with aortic valve disease undergoing TAVR will be enrolled. Clinical follow-up will be conducted in the periprocedural and after TAVR at 1 month, 5 years, and 10 years
  Other Names: Transcatheter aortic valve implantation

SUMMARY:
This registry aims to evaluate the long-term prognosis and valve durability of transcatheter aortic valve replacement (TAVR) in a real-world setting. Baseline characteristics, procedural data, and clinical outcomes will be collected in a prospective and observational manner.

ELIGIBILITY:
Inclusion Criteria:

Patients diagnosed with severe aortic valve regurgitation undergo evaluation by the Heart team and are eligible for TAVR therapy.

2. Patients who understand the purpose of this study, agree to participate in the trial and sign the informed consent form

* 1. Patients with aortic stenosis or aortic valve insufficiency who were evaluated by the Heart team and underwent TAVR therapy
* 2. Patients who understand the purpose of the study, agree to participate in the trial and sign the informed consent form

Exclusion Criteria:

* 1. Patients who cannot provide informed consent
* 2. Patients who are participating in other clinical trials

Min Age: 18 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: Consecutive patients with severe aortic stenosis or valve regurgitation undergo transcatheter aortic valve replacement (TAVR) following evaluation by a cardiac team.
Sampling Method: Non-Probability Sample
Enrollment: 1000 (Estimated)
Dates: Start 2016-01 (Actual); Primary Completion 2025-12 (Estimated); Study Completion 2030-12 (Estimated)

PRIMARY OUTCOMES:
All-casuse mortality | 5 years
  All-casuse mortality including cardiac death and non-cardiac death
Valve-related long-term clinical efficacy | 5 years
  * Freedom from bioprosthetic Valve Failure (defined as: Valve- related mortality OR Aortic valve re-operation/re-intervention OR Stage 3 hemodynamic valve deterioration
  * Freedom from stroke or peripheral embolism (presumably valve-related, after ruling out other non-valve aetiologies)
  * Freedom from VARC Type 2-4 bleeding secondary to or exacerbated by antiplatelet or anticoagulant agents, used specifically for valve-related concerns (e.g. clinically apparent leaflet thrombosis)

SECONDARY OUTCOMES:
Combined early safety and clinical efficacy outcomes | 30 days
  Composed by all-cause mortality, all strokes, life-threatening or fatal bleeding, major vascular, access-related, or cardiac structural complication, acute kidney injury stage 3 or 4, moderate or severe aortic regurgitation, new permanent pacemaker due to procedure-related conduction abnormalities, conduction block and arrhythmia, surgery or intervention related to the device, any hospitalization, myocardial infarction, any other adverse events
Rate of technical success | at exit from procedure room
  * Freedom from mortality
  * Successful access, delivery of the device, and retrieval of the delivery system
  * Correct positioning of a single prosthetic heart valve into the proper anatomical location
  * Freedom from surgery or intervention related to the device or to a major vascular or access-related, or cardiac structural complication
Rate of device success | discharge or 30 days
  * Technical success
  * Freedom from mortality
  * Freedom from surgery or intervention related to the device or to a major vascular or access-related or cardiac structural complication
  * Intended performance of the valve (mean gradient<20mmHg, and less than moderate aortic regurgitation)
Combined clinical efficacy outcomes | 5 years and 10 years
  Combined clinical efficacy outcomes as composed by all-cause mortality (cardiac/non-cardiac), all strokes, any hospitalization
Valve-related long-term clinical efficacy | 10 years
  * Freedom from bioprosthetic Valve Failure (defined as: Valve- related mortality OR Aortic valve re-operation/re-intervention OR Stage 3 hemodynamic valve deterioration
  * Freedom from stroke or peripheral embolism (presumably valve-related, after ruling out other non-valve aetiologies)
  * Freedom from VARC Type 2-4 bleeding secondary to or exacerbated by antiplatelet or anticoagulant agents, used specifically for valve-related concerns (e.g. clinically apparent leaflet thrombosis)

CONTACTS AND LOCATIONS:
Overall Officials: Ling Tao, M.D, Ph.D, Study Chair — Xijing Hospital; Rutao Wang, M.D, Ph.D, Study Chair — Xijing Hospital
Locations (1):
- Xijing Hospital, Xi'an, Shannxi, China